CLINICAL TRIAL: NCT03171779
Title: Impact of Interprofessional Training and Co-ordination on Early Identification and Proactive Approach to End-of-life Situations in the Context of Primary Care
Acronym: SCOP3 quali
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2015_843_0038
Record Dates: First submitted 2017-05-29; First posted 2017-05-31 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Interprofessional Relations; End-of-life Situations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Usual practice
  Interventions: Other: Patients approaching the end of their lives
- IPEM: Interprofessional Training in Early Identification and Multidimensional Evaluation (IPEM) of patients' palliative needs
  Interventions: Other: Patients approaching the end of their lives
- IPEM and PAS: Interprofessional Early Identification Training and Multidimensional Assessment (IPEM) of patients' palliative needs, and to the Early Care Planning (SAP)
  Interventions: Other: Patients approaching the end of their lives

INTERVENTIONS:
Other: Patients approaching the end of their lives — To determine whether the use of simple tools by a primary care team for the early identification of end-of-life patients can improve access to specialized palliative care resources

SUMMARY:
More than 300,000 people die each year in France from a disease that may require palliative care. Nevertheless, only a small proportion of these patients are able to access this care, in particular because of a too late identification.

While several factors may hinder access to specialized palliative care resources, one of the major barriers to the initiation of palliative care, and particularly to the implementation of quality end-of-life care, Remains the failure to recognize that patients with advanced chronic illness are actually approaching the end of their lives.

However, it is now clearly established that early integration of palliative care in the care of people living with a serious, incurable and progressive disease:

* has an impact on the quality (and sometimes the expectation) of life of these people,
* avoids aggressive treatments and unplanned hospitalizations,
* is associated with lower health costs than other end-of-life patients. Primary health care providers have a major role to play in facilitating access to palliative care, but their practice has been hampered in our country by the fragmented and poorly coordinated nature of primary care and Negligible in terms of training. However, they remain the first contact of the patients with the system of care, and are also structuring for the continuation of the patient's journey within the health system.

The first hypothesis is that the work of genuine interprofessional primary care teams in multi-professional health centers (MSPs), coupled with adequate training in the use of simple tools, can contribute to the early identification of patients approaching End of life, to meet their palliative care needs.

However, various European programs (Gold Standards Framework in the UK, NECPAL in Catalonia, RADPAC in the Netherlands) have shown that identification alone is not enough to increase access to specialized palliative care. The second hypothesis is that it must be articulated for this with a training of the professionals to carry out conversations of anticipated planning of the care with their patients.

ELIGIBILITY:
Inclusion Criteria:

* Being a multi-professional health care home (MSP)
* At least one specialized palliative care resource available in the MSP territory (USP, EMSP, palliative care network)

Exclusion Criteria:

* Health centers, group medical practices, clinics
* Less than 3 general practitioners (GPs) and / or absence of nurses (FDI) within the MSP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Being a multi-professional health care home (MSP)
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2015-06-17 (Actual); Primary Completion 2027-10-18 (Estimated); Study Completion 2027-10-18 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who have died from a condition that may require palliative care | 3 years
  Proportion of patients who have died from a condition that may require palliative care

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No